CLINICAL TRIAL: NCT05416970
Title: The Influence of Superimposed Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Lifestyle Changes on Non-alcoholic Fatty Liver Disease Evolution: a Matter of Body Composition
Brief Title: The Influence of SARS-CoV-2 Lifestyle Changes on Non-alcoholic Fatty Liver Disease Evolution
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alessandro Federico, Full Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 15.04-20220010000
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: SARS-CoV-2; non-alcoholic fatty liver disease; Bioelectrical impedance analysis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-alcoholic fatty liver disease affected patients: Patients affected by NAFLD based on clinical, biochemical, imaging and histology, in accordance to CPG diagnostic criteria, continuously followed by the Hepato-gastroenterology Division of the University of Campania Luigi Vanvitelli, between January 2018 and January 2022 were enrolled, after signing an informed consent, in the present study.
  Interventions: Behavioral: SUPERIMPOSED SEVERE ACUTE RESPIRATORY SYNDROME CORONAVIRUS-2 (SARS-CoV-2) LIFESTYLE CHANGES

INTERVENTIONS:
Behavioral: SUPERIMPOSED SEVERE ACUTE RESPIRATORY SYNDROME CORONAVIRUS-2 (SARS-CoV-2) LIFESTYLE CHANGES — To assess the impact of the SARS-CoV-2 spread related lifestyle changes on body composition analysis and metabolic syndrome components worsening as well as hepatocellular carcinoma occurrence.

SUMMARY:
Unhealthy lifestyle represents a key element fueling the non-alcoholic fatty liver disease (NAFLD) onset and worsening. The investigators aimed to evaluate the effects of confinement-related lifestyle changes experienced during the Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) pandemic on NAFLD evolution. A retrospective cohort of NAFLD patients was followed two years before and two years during the pandemic. At three identified time points [baseline (January 2018: T0), intermediate (January 2020: T1), and end of study (January 2022: T2)], anthropometrical, biochemical, nutritional, bioelectrical impedance analysis (BIA) data and non-invasive tools measurements were collected.

DETAILED DESCRIPTION:
The investigators performed a four years retrospective study on a NAFLD cohort from January 2018 to January 2022, dividing the study period in accordance to the beginning of the European SARS-CoV-2 spread in January 2020: two years before the pandemic followed by an equal period during the pandemic. The investigators routinely followed-up the enrolled patients with clinical, biochemical and imaging assessments in accordance with the current CPG and presented the data as mean values of the recordings occurred during the specific period of observation for insulin, fasting plasma glucose (FPG), the homeostatic model assessment for insulin resistance (HOMA-IR), aspartate aminotransferase (AST), alanine aminotransferase (ALT), platelets count (PLT), plasma albumin. Baseline (T0), intermediate (at the end of the pre-pandemic period, January 2020: T1), and end of the study (January 2022 T2) weight, body mass index (BMI), liver stiffness measurement (LSM) and controlled attenuation parameter (CAP), NAFLD fibrosis score (NFS) and multicompartment bioimpedance body composition analysis were also performed. Moreover, a physical activity investigation in terms of hours per week of physical exercise and daily caloric intake were collected by administering a standardized questionnaire. The Alcohol Use Disorders Identification Test (AUDIT-C) questionnaire was also recorded to assess alcohol consumption.

For the entire length of the study, the investigators screened and eventually recorded hepatocellular carcinoma (HCC) occurrence by using ultrasonography assessments in accordance with CPG.

The study primary endpoint was to assess the impact of the SARS-CoV-2 spread related lifestyle changes on body composition analysis and metabolic syndrome components worsening. Secondary endpoint was to assess the impact of the pandemic on HCC occurrence as well as shed light on the pandemic risk factors for HCC onset.

ELIGIBILITY:
Inclusion Criteria:

- NAFLD diagnosis based on clinical, biochemical, imaging and/or histology

Exclusion Criteria:

* diagnosis of inflammatory bowel disease,
* diagnosis of acute kidney disease
* diagnosis of chronic kidney disease
* diagnosis of rheumatoid arthritis
* diagnosis of systemic lupus erythematosus
* diagnosis of other major systemic autoimmune diseases
* diagnosis of tumors
* diagnosis of ongoing infections
* diagnosis of alcohol or drug abuse
* diagnosis of other etiologies of chronic liver damage
* diagnosis of previous HCC
* use of hepatoprotective drugs
* psychological/psychiatric problems that could have invalidate the informed consent.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by NAFLD based on clinical, biochemical, imaging and histology, in accordance to CPG diagnostic criteria, continuously followed by the Hepato-gastroenterology Division of the University of Campania "Luigi Vanvitelli, between January 2018 and January 2022 were enrolled, after signing an informed consent, in the present study.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Changes of body free fat mass | from January 2018 to January 2022
  A multifrequency bioelectrical impedance analysis (BIA) system (InBody, Seoul, Korea) was used to perform the body composition assessment. For the analysis, two electrodes on the right foot and hand were placed. Using the reactance (Xc), resistance (R) and phase angle [arctangent (Xc/R) × (180/π)] the BIA system, thanks to a series of machineries algorithms elaborated the total body water (TBW), the intracellular and extracellular body water (ICW/ECW), the FFM, the FM, body cell mass (BCM) expressed both in percentage and kilograms (Kg), Skeletal-Muscle-Mass (SMM) in Kg. SMM-Index (SMMI) was calculated by dividing the SMM by the square of the height (m2).
Changes of body fat mass | from January 2018 to January 2022
  A multifrequency bioelectrical impedance analysis (BIA) system (InBody, Seoul, Korea) was used to perform the body composition assessment. For the analysis, two electrodes on the right foot and hand were placed. Using the reactance (Xc), resistance (R) and phase angle [arctangent (Xc/R) × (180/π)] the BIA system, thanks to a series of machineries algorithms elaborated the total body water (TBW), the intracellular and extracellular body water (ICW/ECW), the FFM, the FM, body cell mass (BCM) expressed both in percentage and kilograms (Kg), Skeletal-Muscle-Mass (SMM) in Kg. SMM-Index (SMMI) was calculated by dividing the SMM by the square of the height (m2).
Changes of body cell mass | from January 2018 to January 2022
  A multifrequency bioelectrical impedance analysis (BIA) system (InBody, Seoul, Korea) was used to perform the body composition assessment. For the analysis, two electrodes on the right foot and hand were placed. Using the reactance (Xc), resistance (R) and phase angle [arctangent (Xc/R) × (180/π)] the BIA system, thanks to a series of machineries algorithms elaborated the total body water (TBW), the intracellular and extracellular body water (ICW/ECW), the FFM, the FM, body cell mass (BCM) expressed both in percentage and kilograms (Kg), Skeletal-Muscle-Mass (SMM) in Kg. SMM-Index (SMMI) was calculated by dividing the SMM by the square of the height (m2).
Changes of body Skeletal-Muscle-Mass | from January 2018 to January 2022
  A multifrequency bioelectrical impedance analysis (BIA) system (InBody, Seoul, Korea) was used to perform the body composition assessment. For the analysis, two electrodes on the right foot and hand were placed. Using the reactance (Xc), resistance (R) and phase angle [arctangent (Xc/R) × (180/π)] the BIA system, thanks to a series of machineries algorithms elaborated the total body water (TBW), the intracellular and extracellular body water (ICW/ECW), the FFM, the FM, body cell mass (BCM) expressed both in percentage and kilograms (Kg), Skeletal-Muscle-Mass (SMM) in Kg. SMM-Index (SMMI) was calculated by dividing the SMM by the square of the height (m2).
Changes of body SMM-Index | from January 2018 to January 2022
  A multifrequency bioelectrical impedance analysis (BIA) system (InBody, Seoul, Korea) was used to perform the body composition assessment. For the analysis, two electrodes on the right foot and hand were placed. Using the reactance (Xc), resistance (R) and phase angle [arctangent (Xc/R) × (180/π)] the BIA system, thanks to a series of machineries algorithms elaborated the total body water (TBW), the intracellular and extracellular body water (ICW/ECW), the FFM, the FM, body cell mass (BCM) expressed both in percentage and kilograms (Kg), Skeletal-Muscle-Mass (SMM) in Kg. SMM-Index (SMMI) was calculated by dividing the SMM by the square of the height (m2).
Statistically significant worsening of waist/hip ratio | from January 2018 to January 2022
  For the entire length of the study biochemical and clinical parameters were collected comparing the values of pre pandemic period to the pandemic one
Statistically significant worsening of fasting plasma glucose | from January 2018 to January 2022
  For the entire length of the study biochemical and clinical parameters were collected comparing the values of pre pandemic period to the pandemic one
Statistically significant worsening of blood pressure | from January 2018 to January 2022
  For the entire length of the study biochemical and clinical parameters were collected comparing the values of pre pandemic period to the pandemic one
Statistically significant worsening high density lipoprotein | from January 2018 to January 2022
  For the entire length of the study biochemical and clinical parameters were collected comparing the values of pre pandemic period to the pandemic one
Statistically significant worsening triglycerides | from January 2018 to January 2022
  For the entire length of the study biochemical and clinical parameters were collected comparing the values of pre pandemic period to the pandemic one

SECONDARY OUTCOMES:
rate of hepatocellular carcinoma occurrence | from January 2018 to January 2022
  For the entire length of the study the new onset of HCC were recorded comparing the pre pandemic period to the pandemic one

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Federico, Professor, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
All the data that underlie results in a publication are available for the IPD sharing process upon reasonable request to the principal investigator. The access to the data will be granted to Researchers who provide a methodologically sound proposal. Proposals should be directed to alessandro.federico@unicampania.it or marcello.dallio@unicampania.it. To gain access, data requestors will need to sign a data access agreement. Data are available starting 6 months after publication for 10 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication for 10 years
Access Criteria: All the data that support the results of the publication will be shared upon reasonable request by correspondence to alessandro.federico@unicampania.it or marcello.dallio@unicampania.it

REFERENCES:
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Associazione Italiana per lo Studio del Fegato (AISF), Societa Italiana di Diabetologia (SID) and Societa Italiana dell'Obesita (SIO); Members of the guidelines panel; Coordinator; AISF Members; SID Members; SIO Members; Metodologists. Non-alcoholic fatty liver disease in adults 2021: A clinical practice guideline of the Italian Association for the Study of the Liver (AISF), the Italian Society of Diabetology (SID) and the Italian Society of Obesity (SIO). Nutr Metab Cardiovasc Dis. 2022 Jan;32(1):1-16. doi: 10.1016/j.numecd.2021.04.028. Epub 2021 Dec 16. PMID 34924246